CLINICAL TRIAL: NCT04487925
Title: A Randomized Comparison of One Controlled Ovarian Stimulation With Corifollitropin Alfa Versus up to Three Modified Natural Cycles in Expected and Established Poor Responders
Brief Title: Controlled Ovarian Stimulation Versus Modified Natural Cycles in Poor Responders
Acronym: MONACO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-09933
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Reserve; Poor Responders; IVF
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; follitropin beta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Up to 3 modified natural cycles (Active Comparator)
  Interventions: Drug: Up to three modified natural cycles with Follitropin beta.
- Controlled ovarian stimulation (Experimental)
  Interventions: Drug: A single Gonadotropin-Releasing Hormone (GnRH) antagonist corifollitropin alfa (CFA) stimulation

INTERVENTIONS:
Drug: A single Gonadotropin-Releasing Hormone (GnRH) antagonist corifollitropin alfa (CFA) stimulation — CFA will be administered in combination with Follitropin beta.
  Arms: Controlled ovarian stimulation
Drug: Up to three modified natural cycles with Follitropin beta. — Follitropin beta in a low dose will be given.
  Arms: Up to 3 modified natural cycles

SUMMARY:
This is a prospective, randomized, single center, phase 4 controlled trial. The study will compare the efficacy of two different strategies for the management of predicted poor response patients under stimulation for IVF/ICSI: up to three MNC cycles (group 1) versus a single GnRH antagonist CFA (group 2).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (ICF) dated and signed.
* Age ≥18 and <45 years old.
* Body Mass Index (BMI) ≥18.5 Kg/m² and <35 Kg/m².
* Regular menstrual cycles (between 21 and 35 days).
* Two ovaries present.
* Current pregnancy wish.
* Poor responders as defined according to the POSEIDON criteria:

POSEIDON Group 3: patients < 35 years with poor ovarian reserve pre-stimulation parameters (AFC <5 or AMH <1.2 ng/mL); POSEIDON Group 4: patients ≥35 years with poor ovarian reserve pre-stimulation parameters (AFC <5 or AMH <1.2 ng/mL).

Exclusion Criteria:

* Simultaneous participation in another clinical study.
* Untreated and uncontrolled thyroid dysfunction.
* Tumors of the ovary, breast, uterus, pituitary or hypothalamus.
* Abnormal (not menstrual) vaginal bleeding without a known/diagnosed cause.
* Ovarian cysts or enlarged ovaries.
* Malformations of the reproductive organs.
* Current use of oral contraceptives, anti-psychotics, anti-epileptics or chemotherapy.
* Previous antibiotic hypersensitivity reactions (streptomycin and/or neomycin).
* Patients who undergo preimplantation genetic testing (PGT), fertility preservation or oocyte donation.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of good quality blastocysts after CFA stimulation vs. after a first MNC | On fifth day of embryonal development

SECONDARY OUTCOMES:
Number of good quality blastocysts after CFA stimulation vs. after a second or third MNC | On fifth day of embryonal development
The relative number of blastocysts after ART, relative to the number of oocytes | On fifth day of embryonal development
The probability of having at least one blastocyst of good quality after ART | On fifth day of embryonal development

OTHER OUTCOMES:
The probability of having an ongoing pregnancy | 6 to 8 weeks gestational age
The time until ongoing pregnancy | 6 to 8 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Stoop, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No